CLINICAL TRIAL: NCT06690879
Title: ASSESSMENT of UPPER CROSS SYNDROME and CERVICOGENIC HEADACHE AMONG ADDICTIVE SMART PHONE PHYSICAL THERAPY STUDENTS
Brief Title: Assessment of Upper Cross Syndrome and Cervicogenic Headache in Smart Phone User
Status: Completed | Type: Observational
Sponsor: Jilan Adel yousef (Other)
Responsible Party: Sponsor-Investigator, Jilan Adel yousef, doctor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: postural disorder
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Postural; Defect
Keywords: smart phone addiction upper cross syndrome cervicogenic headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- addictive smart phone group: addictive smart phone users with cervicogenic headache
  Interventions: Device: Smartphone application AI Posture Evaluation and Correction System (APECS)
- non addictive smart phone group: non addictive smart phone users not complaining of cervicogenic headache
  Interventions: Device: Smartphone application AI Posture Evaluation and Correction System (APECS)

INTERVENTIONS:
Device: Smartphone application AI Posture Evaluation and Correction System (APECS) — Mobile application APECS v. 6.2.0. is used to assess upper body posture during standing from back side and right side.

SUMMARY:
the purpose of this study was to assess upper cross syndrome and cervicogenic headache between addictive and non- addictive smartphone usage among university physical therapy students.

DETAILED DESCRIPTION:
"Smartphone addiction" is a special type of technological addiction. users are drawn to it Even when there isn't a pressing need to use a smartphone. In a study of 2367 university students in Riyadh, the findings showed that 27.2% of participants used their smartphones for more than eight hours a day. When using a smartphone, a person may stay still for extended periods of time or perform certain movements repeatedly, which puts an excessive amount of static load on the neck and shoulder regions. The most common complaints on smartphones were related to neck pain, with prevalence rates ranging from 17.3% to 67.8%. This is because using a smartphone for extended periods of time with flexed-necked posture increases the activity of the upper trapezius and splenius capitis muscles, which can cause pain in the neck and shoulders. upper crossed syndrome (USC) is muscle imbalance between tightness and weakness in the neck, shoulders, and upper back which is a common postural dysfunction pattern. The main UCS feature is forward head posture (FHP) which is a condition occurs when the head shifts from its usual position and moves forward from the cervical spine. Postural abnormalities associated with UCS include change in the activation of the scapula muscles result in scapular instability and mechanical dysfunction in the neck, which can exacerbate pain in the neck ,upper back and headaches. The International Headache Society (IHS) defines cervicogenic headache (CGH) as a secondary type of headache brought on by abnormalities of the cervical spine or any of the bone, soft tissue, or disc components that make up the cervical spine. A recent study evaluated the frequency of cervicogenic headaches caused by excessive use of smart devices found 56% of students experienced cervicogenic headaches as a result of using smart devices excessively and adopting poor posture. So the aim of this study to assess upper cross syndrome and cervicogenic headache between addictive and non-addictive smartphone usage among university physical therapy students.

ELIGIBILITY:
Inclusion Criteria:

* 1. Asymptomatic students with normal healthy state 2. Age group between 18-24 years 3. Body mass index between (18-24.9). 4. Addictive smart phone users with score over 31 for male and 33 for female students in smart phone addiction scale (Kwon et al., 2013).

  5. Minimum of 25 text messages or emails per day, browsing the Internet and/or playing games for more than one hour a day using their smartphone (Mustafaoglu et al., 2021).
  1. Headache developed in temporal relation to the onset of cervical disorder or appearance of the lesion.
  2. Headache significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion.
  3. Reduced cervical range of motion , and headache was made significantly worse by provocative maneuvers.
  4. Headache abolished following diagnostic blockade of a cervical structure or its nerve supply

     Exclusion Criteria:
* 1. History of Cervical Trauma or Surgery (Jung et al., 2016). 2. Neck, shoulder, upper back, lower back, elbow, or wrist-hand musculoskeletal trauma (Lee et al., 2015).

  3. Congenital deformities 4. Serious surgical or neurological diseases 5. Limb injuries 6. Involvement in a formal physical activity program 7. Cervical Spondylosis. 8. Cervical Radiculopathy (Pathan et al., 2021). 9. Shoulder, neck, and back muscle injuries in the past month (Daniel et al., 2022).

  10. Idiopathic spinal deformity (Elnahhas et al., 2018).

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: smart phone users from faculty of physical therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
upper cross syndrome angles assessment in degrees | 3 monthes
  cranio-vertebral angle ,rounded shoulder and Thoracic kyphosis angles .

SECONDARY OUTCOMES:
cervical range of motion in degrees and flexion rotation test in degree | 3 months
  features of cervicogenic headache

CONTACTS AND LOCATIONS:
Overall Officials: enas fawzy, professor, Study Director — professor of physical therapy for orthopedic diseases
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trovato B, Roggio F, Sortino M, Zanghi M, Petrigna L, Giuffrida R, Musumeci G. Postural Evaluation in Young Healthy Adults through a Digital and Reproducible Method. J Funct Morphol Kinesiol. 2022 Oct 28;7(4):98. doi: 10.3390/jfmk7040098. PMID 36412760
- [Background] Stenneberg MS, Busstra H, Eskes M, van Trijffel E, Cattrysse E, Scholten-Peeters GGM, de Bie RA. Concurrent validity and interrater reliability of a new smartphone application to assess 3D active cervical range of motion in patients with neck pain. Musculoskelet Sci Pract. 2018 Apr;34:59-65. doi: 10.1016/j.msksp.2017.12.006. Epub 2017 Dec 16. PMID 29328979
- [Background] Kwon M, Lee JY, Won WY, Park JW, Min JA, Hahn C, Gu X, Choi JH, Kim DJ. Development and validation of a smartphone addiction scale (SAS). PLoS One. 2013;8(2):e56936. doi: 10.1371/journal.pone.0056936. Epub 2013 Feb 27. PMID 23468893
- [Background] Alageel AA, Alyahya RA, A Bahatheq Y, Alzunaydi NA, Alghamdi RA, Alrahili NM, McIntyre RS, Iacobucci M. Smartphone addiction and associated factors among postgraduate students in an Arabic sample: a cross-sectional study. BMC Psychiatry. 2021 Jun 10;21(1):302. doi: 10.1186/s12888-021-03285-0. PMID 34112121